CLINICAL TRIAL: NCT04426305
Title: Community Health Workers Against COVID19 Tackling Psychosocial Suffering Due to Physical Distancing
Brief Title: Community Health Workers Against COVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BC-07744.
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2020-05

CONDITIONS: Covid 19; Social Isolation; Mental Health Impairment
Keywords: Community health workers; randomized controlled trial; psychosocial impairment
MeSH Terms: conditions — COVID-19; Social Isolation

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): psychosocial support
  Interventions: Other: community health worker support
- control arm (Active Comparator): care as usual
  Interventions: Other: care as usual

INTERVENTIONS:
Other: community health worker support — usual care by professional primary care providers + emotional support by trained community health worker
  Arms: Intervention arm
Other: care as usual — care as usual is provided by professional primary care provider
  Arms: control arm

SUMMARY:
Randomized controlled trial among patients from family practices at risk of psychosocial suffering due to social distancing measures. Patients from the intervention group receive support from community health workers. contacted at least 8 times by community health workers. Evolution of psychosocial wellbeing is evaluated by questionnaires at time 0 and after 6 weeks of intervention. Psychosocial outcomes are compared between control and intervention groups. Process evaluation will be done through in-depth interviews.

DETAILED DESCRIPTION:
Patients vulnerable for psychosocial suffering due to social distancing measures are recruited by family practitioners in the City of Ghent. The recruited patients are randomly selected into a control and intervention group. Based on the validated Promis instruments, all participants are interviewed face to face on their mental and social health at time 0 and after 6 weeks of intervention. Patients from the intervention group are contacted by Community health workers after the first interview. Community health workers offer emotional support to the patients through at least 8 contacts over 6 weeks. The control group receive care as usual and are offered support by community health workers after the second interview. In depth interviews (qualitative study) will be conducted among community health workers and patients after finalizing the post-intervention questionnaires.

Research questions: What are the psychosocial consequences of social distancing for at-risk groups? Can community health workers reduce the psychosocial impact of physical distancing measures isolation?

Relevance: Understanding community-based psychosocial support for vulnerable people during and after health crises.

Keywords: Community health workers, psychosocial, health crises

ELIGIBILITY:
Inclusion Criteria:

* patients recruited by family practitioners based on anticipated psychosocial impact of physical distancing measures

Exclusion Criteria:

* Patients with severe psychiatric diseases (psychosis, severe depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported Emotional Support (based on the PROMIS® Emotional Support instrument) | change from baseline at 6 weeks
  The PROMIS Emotional Support questionnaire assesses perceived feelings of being cared for and valued as a person;
Change in patient-reported Social Isolation (based on the PROMIS® Emotional Support instrument) | change from baseline at 6 weeks
  The PROMIS Social Isolation questionnaire assesses perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others.
Change in patient-reported Ability to participate in social roles and activities (based on the PROMIS® ability to participate in social roles and activities instrument) | change from baseline at 6 weeks
  The PROMIS adult Ability to Participate in Social Roles and Activities questionnaire assesses the perceived ability to perform one's usual social roles and activities.
Change in patient-reported anxiety (based on the PROMIS® anxiety instrument) | change from baseline at 6 weeks
  The PROMIS Anxiety questionnaire assesses self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health and Primary Care, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR